CLINICAL TRIAL: NCT01498926
Title: A Randomised, Single Centre, Two-period, Cross-over, Glucose Clamp Trial to Test for Bioequivalence Between Two Insulin Detemir Formulations Containing Mannitol and Glycerol as Isotonic Agents Respectively, in Healthy Subjects
Brief Title: Comparison of Two Insulin Detemir Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1685; 2005-002481-11 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycerol (Experimental)
  Interventions: Drug: insulin detemir
- Mannitol (Active Comparator)
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Single dose containing mannitol as isotonic agent. Administered subcutaneously (s.c., under the skin)
  Arms: Mannitol
Drug: insulin detemir — Single dose containing glycerol as isotonic agent. Administered subcutaneously (s.c., under the skin)
  Arms: Glycerol

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare two formulations of insulin detemir containing an isotonic agent in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body mass index (BMI) between 18 and 27 kg/m^2, inclusive
* Non-smoker
* Fasting plasma glucose maximum 6 mmol/L

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Previous participation in this trial
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (intrauterine device (IUD) that has been in place for at least 3 months, sterilisation, the oral contraceptive pill (which should have been taken without difficulty for at least 3 months) or an approved hormonal implant)
* The receipt of any investigational drug within the last 3 months prior to this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2005-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin detemir concentration curve
Maximum serum insulin concentration

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve
Time to maximum serum insulin concentration
Terminal serum insulin half life
Area under the serum insulin detemir concentration curve
Maximum glucose infusion rate
Time to maximum glucose infusion rate
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Manchester, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com